CLINICAL TRIAL: NCT06442085
Title: Immersive Virtual Reality Versus Mannequin-based Simulation Training for Trauma Resuscitation: a Randomized Controlled Non-inferiority Trial
Brief Title: Virtual Reality Training for Trauma Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riga Stradins University (Other)
Responsible Party: Principal Investigator, Ainars Stepens, Lead researcher in Institute of Public Health, Riga Stradins University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RigaStradinsU
Record Dates: First submitted 2024-05-20; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Virtual Reality
Keywords: Virtual reality; trauma; simulation-based education; resuscitation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This was a prospective, single-center, randomized, controlled, non-inferiority, simulation-based trial comparing the use of virtual reality simulation vs. mannequin based simulation in a simulated trauma scenario.
Who Masked: Outcomes Assessor
Masking Description: All assessments of the student performances were recorded either by video camera (mannequin based simulation) or screen capture (virtual reality simulation). All videos were assessed by two blinded raters independently. In order to maintain consistency, virtual reality recordings were also scored manually by the raters, instead of the automated Trauma Simulator built-in tool. The video data were stored for the reviews and deleted afterwards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical students - volunteers receiving mannequin based simulation training (Active Comparator): volunteers receiving mannequin based simulation training (control), then assessed for primary outcome, analyzed for primary outcome.
  Interventions: Other: Teaching of trauma resuscitation by using mannequin based simulation
- Medical students - volunteers receiving virtual reality simulation training (Experimental): volunteers receiving virtual reality simulation training (intervention), then assessed for primary outcome, analyzed for primary outcome.
  Interventions: Other: Teaching of trauma resuscitation by using virtual reality simulation

INTERVENTIONS:
Other: Teaching of trauma resuscitation by using virtual reality simulation — The intervention was teaching of trauma resuscitation by using VRS. Following welcome and a video lecture by Advance Trauma Life Support certified physician, the intervention group participants were orientated (15 minutes) to the VRS environment, head-mounted display (Oculus Rift S or Oculus Quest, Oculus, USA) and hand controllers by playing game First Steps (Oculus, USA). Then the participants were training by using the "Internal Hemorrhage" scenario in Trauma Simulator.
  Arms: Medical students - volunteers receiving virtual reality simulation training
Other: Teaching of trauma resuscitation by using mannequin based simulation — Volunteers were trained in groups of three or four by using mannequin-based rapid cycle deliberate practice simulation facilitated by a critical care physician. Next, the volunteers had 50 min training of the same trauma scenario as the intervention group. The simulation facility was set-up as close as possible to the virtual reality environment.
  Arms: Medical students - volunteers receiving mannequin based simulation training

SUMMARY:
This study individual training with an immersive virtual reality Trauma Simulator was compared to live mannequin-based simulation training in a facilitated group. The results showed that virtual reality simulator led to non-inferior effects on trauma resuscitation skills to mannequin-based simulation. Trauma Simulator had good usability, was well received by the participants, and had minimal adverse effects.

DETAILED DESCRIPTION:
Background: Despite its high potential, the effect of immersive virtual reality simulation (VRS) in trauma resuscitation training has not been studied. The aim of this study was to test the hypothesis that VRS is non-inferior to mannequin-based simulation (MBS) in trauma resuscitation training.

Methods: In a single-center, randomized controlled non-inferiority trial, we compared individual training with an immersive virtual reality Trauma Simulator to live MBS training in a facilitated group. The primary outcome was the Trauma Score (ranging from 55 (worse) to 177 (best outcome)) during the MBS assessment. The secondary outcomes were the Trauma Score VRS assessment, System Usability Scale (ranging from 0 (worse) -100 (best outcome)), and Simulation Sickness Questionnaire (ranging from 0 (worse) to 235.62 (best outcome)).

ELIGIBILITY:
Inclusion Criteria: fluency in English. Exclusion Criteria: history of motion sickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Trauma Score | Within a Day
  The primary outcome of the study is Trauma Score (range 55 (worst) to 177(best outcome) during an individual assessment in a mannequin-based simulation environment. The assessment was based on the video recordings analyzing students during performing in the scenario. The Trauma Score is an assessment tool developed by military emergency medicine experts for the Trauma Simulator.

SECONDARY OUTCOMES:
Trauma Score in VRS | Within a VR session (less than 10minutes per person)
  Trauma Score in the VRS environment served as a secondary outcome. System Usability Scale: a 10-item questionnaire (range 0-100, where 0 is the worst, 100 the best performance) was used to assess usability of Trauma Simulator.
Pre- and Post-Surveys | Within a Day
  The students will receive pre and post surveys. The surveys are structured to evaluate students' experience before and after the training. As a reference, the evaluation tools are made, based on Bangor et al., 2009. A custom, six-question survey (5-point Likert scale) was used to assess the perception of Virtual Reality simulation before and after the study. Presence of cybersickness was evaluated by using Simulation Sickness Questionnaire (SSQ).15 SSQ assesses 16 symptoms of motion sickness in three domains: nausea (7 symptoms), disorientation (7 symptoms), and oculomotor effects (7 symptoms). Each symptom is self-reported as none (0), slight (1), moderate (2), and severe (3). Total Severity score is calculated as the sum of individual symptom scores in each domain multiplied by 3.74 in accordance with Kennedy et al. (1993), thus the final score ranges from 0 (worst) to 235.62 (best outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Ainars Stepens, PhD, MD, Principal Investigator — Institute of Public Health, Riga Stradiņš University
Locations (1):
- Medical Education Technology Centre of Riga Stradins University, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No
Participants were volunteers. Their data has been protected by General data protection regulation (GDPR). The anonymized Trauma Score of each participant group is available upon request.

REFERENCES:
- [Background] Bangor A, Kortum P: Determining what individual SUS scores mean: adding an adjective rating scale. Journal of Usability Studies. 2009;4:114-123.
- [Background] Kennedy RS, Lane NE, Berbaum KS, Lilienthal MG: Simulator Sickness Questionnaire: an enhanced method for quantifying simulator sickness. The International Journal of Aviation Psychology. 1993;3:203-220.
- See also: POWER (SAMPLE SIZE) CALCULATORS' — https://www.sealedenvelope.com/power/continuous-noninferior/
- See also: G. C. Urbaniak and S. Plous, 'RESEARCH RANDOMIZER - RANDOM SAMPLING AND RANDOM ASSIGNMENT MADE EASY! — https://www.randomizer.org